CLINICAL TRIAL: NCT07289295
Title: Prospective Clinical Study to Evaluate the Safety and Efficacy of Versius in Robot-Assisted Total Hysterectomy
Brief Title: Versius Gynecology Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CMR Surgical Ltd (Industry)
Collaborators: Uniwersyteckie Centrum Kliniczne im. prof. K. Gibińskego Śląskiego Uniwersytetu Medycznego w Katowicach (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA-00574
Record Dates: First submitted 2025-07-30; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Robotic Assisted Hysterectomy and/or Salpingo-oophorectomy
Keywords: Versius; robotic surgery; hysterectomy; salpingo-oophrectomy; gynecology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Surgery with Versius (Experimental)
  Interventions: Device: Versius Surgical System

INTERVENTIONS:
Device: Versius Surgical System — Modular robotic system intended to assist in the accurate control of its surgical endoscopic instruments across a range of surgical procedures

SUMMARY:
The objective of this clinical trial is to expand the clinical evaluation of the safety and efficacy of Versius in gynaecology procedures of total robotic assisted hysterectomy and/or salpingo-oophorectomy

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged 22 years or above, who provided written informed consent to participate in the study.
2. Patient deemed suitable for minimally invasive total hysterectomy and/or Salpingo-Oophorectomy, for benign condition.
3. Patient with BMI ≤40.

Exclusion Criteria:

1. Patient unwilling to provide informed consent.
2. Medical contraindication for general anaesthesia or minimally invasive procedure.
3. Oncological cases, patient undergoing surgery or treatment for malignant disease.
4. Clinically assessed Uterus size of > 14 pregnancy weeks (Estimated as > 14-15 cm longitudinal diameter).
5. Patient participation in an interventional clinical study that could impact primary outcomes results.
6. Patient who falls into American Society of Anaesthesiologists (ASA) Class IV or above (Appendix A).
7. Uncontrolled hypertension, uncontrolled diabetes mellitus, or kidney failure.

Min Age: 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Success rate | Day of surgery
  Rate of successful completion of robotic assisted surgery without unplanned conversion to other laparoscopic or open surgery.
Serious Adverse Event rate | Up to 30 days post procedure
  Rate of total serious adverse events

SECONDARY OUTCOMES:
Operative time | Day of surgery
  Surgical time from skin incision to skin closure
Estimated blood loss | Day of surgery
  Amount of blood estimated to be lost during surgery (in mL)
Intra-operative complications | Day of surgery
  Complications that occur during surgery
Blood transfusions | Up to post-surgical discharge, i.e. the date when patient is considered sufficiently recovered from surgery to leave hospital, expected to be at most up to 1 month after date of surgery, typically within a few days
  Need for blood transfusion during or after surgery as well as amount transfused
Unplanned instrument use | Day of surgery
  Whether unplanned use of non-Versius laparoscopic instruments during surgery occurs as well as at what surgical step
Device deficiencies | Day of surgery
  Any device deficiencies of Versius during surgery
Reoperation within 24 hours | 24 hours post-surgery
  Need for reoperation after initial surgery
Length of hospital stay | Up to post-surgical discharge, i.e. the date when patient is considered sufficiently recovered from surgery to leave hospital, expected to be at most up to 1 month after date of surgery, typically within a few days
  Hospital stay in days from day of surgery until discharge
Adverse events | Up to 30 days post-surgery
  Rate of adverse events
Readmission | Up to 30 days post-surgery
  Hospital readmission after post-surgical discharge
Reoperation within 30 days | Up to 30 days post-surgery
  Need for reoperation as a result of interventional surgery itself or the indication for surgery
Mortality rate | Up to 30 days post-surgery
Vaginal vault healing | 42 days post-surgery
  Vaginal vault healing as anticipated for patients that had total laparoscopic hysterectomy

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Nowosielski, MD, Principal Investigator — Uniwersyteckie Centrum Kliniczne im. prof. K. Gibińskego Śląskiego Uniwersytetu Medycznego w Katowicach
Locations (1):
- Uniwersyteckie Centrum Kliniczne im. prof. K. Gibińskego Śląskiego Uniwersytetu Medycznego w Katowicach, Katowice, Poland

IPD SHARING:
Plan to Share IPD: No